CLINICAL TRIAL: NCT02104986
Title: A Multicenter Study to Evaluate a Risk-adapted Strategy for Treatment of Extra Cranial Non Seminomateous Malignant Germ Cell Tumour in Children and Adolescent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TGM 2013-NS
Record Dates: First submitted 2014-03-27; First posted 2014-04-07 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Extra Cranial Non Seminomateous Malignant Germ Cell Tumour
Keywords: non seminomateous malignant germ cell tumour (NSMGCT); Dose De-escalation; Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3 courses of Velbe-Bleomycin-Cisplatin (Experimental): 3 VBP (Velbe-Bleomycin-Cisplatin) Risk-adapted strategy - reduction of the number of chemotherapy courses
  Interventions: Drug: Velbe-Bleomycin-Cisplatin
- 4 courses of Velbe-Bleomycin-Cisplatin (Experimental): 4 VBP (Velbe-Bleomycin-Cisplatin) Risk-adapted strategy - reduction of the number of chemotherapy courses
  Interventions: Drug: Velbe-Bleomycin-Cisplatin
- 3 courses Vepeside-ifosfamide-Cisplatin (Experimental): 3 VIP (Vepeside-ifosfamide-Cisplatin) Risk-adapted strategy - reduction of the number of chemotherapy courses
  Interventions: Drug: Vepeside-ifosfamide-Cisplatin
- 4 courses Vepeside-ifosfamide-Cisplatin (Experimental): 4 VIP (Vepeside-ifosfamide-Cisplatin) Risk-adapted strategy - reduction of the number of chemotherapy courses
  Interventions: Drug: Vepeside-ifosfamide-Cisplatin

INTERVENTIONS:
Drug: Velbe-Bleomycin-Cisplatin — Limitation of the number of chemotherapy courses (≤ 4) after the achievement of a clinical and biological response in NSMGCT patients treated with cisplatin-based chemotherapy, in order to reduce treatment long-term effects
  Other Names: Desescalation
  Arms: 3 courses of Velbe-Bleomycin-Cisplatin; 4 courses of Velbe-Bleomycin-Cisplatin
Drug: Vepeside-ifosfamide-Cisplatin
  Arms: 3 courses Vepeside-ifosfamide-Cisplatin; 4 courses Vepeside-ifosfamide-Cisplatin

SUMMARY:
The main objective is to assess the benefit-risk ratio of a risk-adapted strategy for treatment of extra cranial NSMGCT in children and adolescent.

DETAILED DESCRIPTION:
Two different situations will be considered:

* in NSMGCT patients treated with cisplatin-based chemotherapy, the objective is to maintain a 2-year progression-free survival rate >80% despite a limitation of the number of course of chemotherapy (≤4) after the achievement of a clinical and biological response (primary endpoint);
* in children over 10 years with testicular or extragonadal NSMGCT, the objective is to improve the overall survival by systematically classifying the patients in high-risk group to allow a dose intensification.

ELIGIBILITY:
Inclusion Criteria:

* Extra cranial non seminomateous malignant germ cell tumour (NSMGCT) except pure immature teratoma.
* Age ≤ 18 years.
* Affiliation with a social security scheme.
* Signed informed consent by parents
* Effective contraception during the study if relevant .

Exclusion Criteria:

* Previous chemotherapy
* Contraindications to study treatments
* Patient who cannot follow medical surveillance due to geographical, social, or psychological reasons
* Pregnant and breast feeding women

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 24 months

SECONDARY OUTCOMES:
Overall survival | Within 10 years after the first inclusion, from the date of inclusion to the date of death due to any cause
complete remission rate after 1st line treatment (chemotherapy and surgery) | 3 weeks after the end of treatment (CT + surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Cécile CONTER, MD, Principal Investigator — Centre Léon Bérard, Lyon, FRANCE
Locations (27):
- France (27):
  - CHU, Amiens
  - CHU, Angers
  - CHRU, Besançon
  - CHU, Bordeaux
  - Chu Morvan, Brest
  - CHU, Caen
  - Chu Estaing, Clermont-Ferrand
  - CHU, Dijon
  - Centre Oscar Lambret, Lille
  - CHU, Limoges
  - Hopital de La Timone, Marseille
  - CHU, Montpellier
  - CHU, Nancy
  - CHU, Nantes
  - CHU, Nice
  - Institut Curie, Paris
  - Hopital Trousseau, Paris
  - CHU, Poitiers
  - CHU, Reims
  - CHU, Rennes
  - CHU, Rouen
  - Hopital Felix Guyon, Saint-Denis
  - CHRU, Saint-Etienne
  - CHRU, Strasbourg
  - CHU, Toulouse
  - CHRU, Tours
  - Institut Gustave Roussy, Villejuif